CLINICAL TRIAL: NCT01572779
Title: A Multicentre, Cluster Randomised, Placebo-controlled, Open-label Pilot Study of Back Strain Monitor (BSM) With Feedback Compared With the BSM Without Feedback in Subjects With Moderate Lower Back Pain.
Brief Title: A Study to Investigate the Effect of a New Postural Bio-feedback Device on Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pro-Active Medical Pty Ltd (Industry)
Collaborators: Department of Business and Innovation, Victoria, Australia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ProA-BSM-001
Record Dates: First submitted 2011-06-07; First posted 2012-04-06 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Low Back Pain
Keywords: dorsavi; vimove; biofeedback; objective movement data; back pain
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): BSM device with bio-feedback
  Interventions: Device: BSM device with bio-feedback
- Control (Placebo Comparator): The BSM device without feed-back
  Interventions: Device: BSM device with no bio-feedback

INTERVENTIONS:
Device: BSM device with bio-feedback — A postural bio-feedback device worn by subjects for 4-10hours a day for 6 days spread across 6 weeks for the sub acute low back pain group and for 8 days spread across 10 weeks for the chronic group. The device records movement and muscle activity data relating to the lower back. Bio-feedback is delivered to the subject as an audible tone, visual cue or vibration and aims to prompt the subject to alter their posture or position in line with recommendations given by the treating practitioner. Four small sensors are adhered to the lower back and send data wirelessly to a data logger carried in the pocket by the subject (the size of a small mobile phone).
  Other Names: ViMove
  Arms: Intervention
Device: BSM device with no bio-feedback — The BSM device is worn as a placebo with no bio-feedback given to the subject. The subjects in the control group wear the device for 4-10 hours a day for 6 days spread across 6 weeks for the sub acute low back pain group and for 8 days spread across 10 weeks for the chronic group.
  Other Names: ViMove with no Feedback
  Arms: Control

SUMMARY:
A postural bio-feedback device worn by subjects for 4-10 hours a day for 6 days spread across 6 weeks for the sub acute low back pain group and for 8 days spread across 10 weeks for the chronic group. The device records movement and muscle activity data relating to the lower back. Bio-feedback is delivered to the subject as an audible tone, visual cue or vibration and aims to prompt the subject to alter their posture or position in line with recommendations given by the treating practitioner. Four small sensors are adhered to the lower back and send data wirelessly to a data logger carried in the pocket by the subject (the size of a small mobile phone).

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides informed consent
2. Age between 18 and 65 years of age
3. At least moderate intensity low back pain (LBP) and/or back related leg pain, as defined by a QVAS score > 3 (Carragee, Spine 2000).
4. Initial QVAS score of > 3 out of 10
5. Subjects must be assessed by the practitioner as Sub Acute (3 to 12 weeks post onset of low back pain (LBP) or Chronic (> 12 weeks post onset of low back pain (LBP).

Exclusion Criteria:

1. Lower back surgery within previous twelve (12) months.
2. Females who are pregnant.
3. Subjects with a severe hearing impairment.
4. Evidence of non mechanical contributing cause for lower back pain e.g. neoplasm, infection, fracture, inflammatory disorder.
5. Preceding chronic neurological changes (Sub Acute group only).
6. Implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator)
7. Nerve block, spinal injection or anesthetic procedure for the treatment of lower back pain within 12 months of the study.
8. Significant medical abnormalities or conditions that in the opinion of the Practitioner would interfere either with the ability to complete the study or the evaluation of the investigational device's safety and efficacy.
9. Recent history of a significant medical-surgical intervention that in the judgment of the Practitioner would interfere either with the ability to complete the study or the evaluation of the investigative device's safety and efficacy.
10. Known allergic skin reaction to tapes and plasters.
11. Subject who is currently enrolled in an investigational drug or device study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionaire (RMDQ-23) | over 12 months
  Functional Outcome measure
Patient Specific Functional Scale (PSFS) | over 12 months
  Functional Outcome Measure
Quadruple Visual Analogue Scale (QVAS) | over 12 months
  Pain Scale

SECONDARY OUTCOMES:
The change over time from baseline in the range of movement, recorded by the device. Measured in degrees of movement in the three anatomical planes. | over 12 months
  Functional Outcome Measure

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jensen, MB BS FAFMM, Principal Investigator — Stanlake Specialist Centre; Adrian Jury, MD, Principal Investigator — Myers Street Family Medical; Joe Garra, MD, Principal Investigator — The Clinic Werribee; Peter Braun, MD, Principal Investigator — Stanlake Specialist Centre; Robert Laird, Principal Investigator — Austin Hospital Pysiotherapy Outpatients
Locations (9):
- Australia (9):
  - Metro Spinal Clinic, Caulfield, Victoria
  - Stanlake Specialist Centre, Footscray, Victoria
  - Myers Street Family Medical, Geelong, Victoria
  - Peak Musculoskeletal, Hampton, Victoria
  - Austin Hopsital, Heidelberg, Victoria
  - Olympic Park Sports Medicine Centre, Melbourne, Victoria
  - Epworth Hospital Richmond, Richmond, Victoria
  - Bounce Health Group, Ringwood, Victoria
  - The Clinic Werribee, Werribee, Victoria

REFERENCES:
- [Derived] Kent P, Laird R, Haines T. The effect of changing movement and posture using motion-sensor biofeedback, versus guidelines-based care, on the clinical outcomes of people with sub-acute or chronic low back pain-a multicentre, cluster-randomised, placebo-controlled, pilot trial. BMC Musculoskelet Disord. 2015 May 29;16:131. doi: 10.1186/s12891-015-0591-5. PMID 26022102
- See also: device description — http://www.dorsavi.com/